CLINICAL TRIAL: NCT01999933
Title: Clinical Study on Docetaxel Plus Cisplatin(TP) Regimen Combined With Postoperative Radiotherapy for Stage Ia2- IIb Cervical Cancer
Brief Title: Evaluation of Postoperative Radiotherapy and Concurrent Chemotherapy Effectiveness in Cervical Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mei Shi (Other)
Responsible Party: Sponsor-Investigator, Mei Shi, Director and Professor of Department of Radiation Oncology, Xijing Hospital, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJFL-201309-CCPOSTOP
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Cervical Cancer; Toxicity Due to Radiotherapy
Keywords: Cervical cancer; postoperative risk factor; treatment
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiation; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CCRT with cisplatin(DDP) weekly (Active Comparator): concurrent chemotherapy: cisplatin（DDP） weekly, 40mg/m2, begin with radiation
  Interventions: Radiation: Radiation; Drug: cisplatin（DDP） weekly
- CCRT with TP (Experimental): concurrent TP tri-weekly, docetaxel plus cisplatin tri-weekly (75mg/m2), begin with radiation
  Interventions: Radiation: Radiation; Drug: docetaxel plus cisplatin
- concurrent and adjuvant TP (Experimental): 2 cycles of concurrent TP, docetaxel plus cisplatin tri-weekly (75mg/m2),begin with radiation; and 4 cycles of adjuvant TP, the same regimen, after radiation
  Interventions: Radiation: Radiation; Drug: docetaxel plus cisplatin

INTERVENTIONS:
Radiation: Radiation — Arm1, Arm2 and Arm3 patients should received the whole pelvic radiation.
Drug: cisplatin（DDP） weekly — concurrent chemotherapy with cisplatin（DDP） weekly(40mg/m2),begin with radiation
  Arms: CCRT with cisplatin(DDP) weekly
Drug: docetaxel plus cisplatin — concurrent docetaxel plus cisplatin tri-weekly (75mg/m2),2 cycles, begin with radiation
  Arms: CCRT with TP; concurrent and adjuvant TP
Drug: docetaxel plus cisplatin — adjuvant chemotherapy with docetaxel plus cisplatin tri-weekly (75mg/m2), 4 cycles after radiation
  Arms: concurrent and adjuvant TP

SUMMARY:
The present study is a randomized, control, phase II/III study of early stage (FIGO Ia2-IIb) cervical cancer after radical hysterectomy in Northwest China treated with radiotherapy or concurrent chemoradiotherapy based on the surgical-pathological risk factors. All the patients received whole pelvis radiation and were divided into three groups according to adjuvant chemotherapy: concurrent chemotherapy with cisplatin weekly (40mg/m2) , concurrent chemotherapy with docetaxel plus cisplatin tri-weekly (75mg/m2), or concurrent and adjuvant chemotherapy with docetaxel plus cisplatin tri-weekly (75mg/m2). The effectiveness, and side effects will be evaluated according to Standard WHO response criteria, and NCI common toxicity criteria for adverse events(NCI-CTC-AE) V3.0.

DETAILED DESCRIPTION:
To the cervical cancer patient who accepted radical hysterectomy, whether the adjuvant therapy should be received or the method of adjuvant therapy are determined by the postoperative pathology. In the traditional opinion, the postoperative risk factors were divided into two groups: intermediate risk factors, including large tumor size, deep stromal invasion and lymphovascular space invasion, and high risk factors, including non-squamous cell carcinoma, marginal positive, parametric invasion and pelvic lymph node(LN) metastasis. Patients with intermediate risk factors should accepted adjuvant radiotherapy only and who with high risk factors should received adjuvant concurrent chemoradiotherapy. Cisplatin weekly(40mg/m2) was the standard regimen of concurrent chemotherapy. However, we retrospectively analyzed 801 cervical cancer patients with postoperative radiotherapy and found that distant metastasis was the main cause of current treatment failure(84.5%), which suggested the current regimen of chemotherapy was insufficient and might be strengthened in future.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 70 Years
* Histologically proven cervical cancer, FIGO stage Ia2-IIb,and no previous chemotherapy and radiotherapy
* Accepted radical hysterectomy 3-4 weeks before
* Karnofsky score >70
* Postoperative pathology with following risk factors: Non-squamous cell carcinoma, deep stromal invasion, lymphovascular space invasion, marginal positive, parametria invasion, large tumor size (tumor diameter>4cm) or pelvic LN metastasis. Patients with pelvic LN metastasis and combination of any two or more risk factors mentioned above were included.
* Examination results showed no radiation or chemotherapy contraindication
* Willing to accept treatment
* Ability to comply with trial requirements

Exclusion Criteria:

* Postoperative residual
* Postoperative recurrence or metastasis
* Without lymph node dissection
* Postoperative pathology showed aortic lymph node metastasis
* Examination results showed radiotherapy contraindications
* No indications for radiotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5-years

SECONDARY OUTCOMES:
disease-free survival | 5 years
acute adverse events | 3 months
chronic adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mei Shi, MD, Principal Investigator — department of radiation oncology
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China